CLINICAL TRIAL: NCT01183624
Title: A Multi-Center, Randomized, Double-Blind, Parallel, Placebo Control Study of a Traditional Chinese Medicine Topical Analgesic Patch in the Treatment of Osteoarthritis of the Knee
Brief Title: A Controlled Study of an Herbal Topical Patch in Treating Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCTPAI3001
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Pain; Herbal medicine; Topical administration
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Patch (Experimental): Herbal Patch
  Interventions: Other: Herbal Patch
- Control Patch (Placebo Comparator): Placebo Patch
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Other: Herbal Patch — 1 herbal patch applied for approximately 8 hours per day for 14 days
  Other Names: Traditional Chinese Medicine Topical Analgesic Patch
  Arms: Experimental Patch
Other: Placebo Patch — Control patch with no herbal ingredients
  Other Names: Not a marketed product
  Arms: Control Patch

SUMMARY:
An evaluation of the safety and efficacy of an herbal patch in treating osteoarthritis pain of the right or left knee.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel-group, placebo-controlled study of herbal patch in subjects with OA knee pain. The overall objective of this study is to evaluate the efficacy and safety of the patch in relieving OA knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 40 and 70 years of age
* Medically cleared to participate by a site affiliated physician following a physical
* History of, or current diagnosis of, OA of the knee
* Evidence of idiopathic OA of at least one knee
* Subject Assessment of OA pain in target knee 40 - 75 mm (on the 100 mm VAS inclusive) in the index knee, on the WOMAC Pain composite subscale at Visit 1
* Subject Assessment of OA pain in non-index knee (if applicable) is ≤ 20mm
* Subject Global Assessment of OA Condition (5 pt categorical scale, 1 = very good to 5 = very poor) of grade 3-5 (i.e. fair, poor or very poor)
* Evidence of idiopathic OA of at least one knee as defined by the American College of Rheumatology Classification (ACR) of OA of the Knee

Exclusion Criteria:

* Grade 1 or Grade 4 severity of the index knee based on the Kellgren and Lawrence radiographic criteria
* Pain greater than 20 mm on the VAS in the non-index knee (either at rest or with movement)
* Prior injection or arthroscopy of study knee within 3 months
* Crystalline-induced synovitis (e.g. gout, pseudo gout, nonsteroid arthritis, hydroxyapatite deposit), acute inflammatory arthritis, rheumatoid arthritis, psoriatic arthritis, septic arthritis, fibromyalgia, systemic lupus, erythematosus collagen vascular disease or other types of inflammatory arthritis in the index knee
* Pain in either knee is of neurological origin
* An injury or surgery to the same body region within the prior 6 months or a lifetime history of 3 or more injuries/surgeries to the injured body region
* Signs of clinically important active inflammation of the study knee joint including redness, warmth, and/or a large, bulging effusion with the loss of normal contour at the screening and/or baseline visits
* Other criteria that - in the opinion of the investigator - may jeopardize the safety of the subject or the study results.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pain Score | Day 7
  The WOMAC (Western Ontario and McMaster Universities Index of Osteoarthritis) Pain Subscale Score

SECONDARY OUTCOMES:
Subject Assessment | Day 3
  Subject Global Assessment of Response to Treatment: WOMAC Physical Function Subscale and Subject Global Assessment of OA Condition
Subject Assessment | Day 7
  Subject Global Assessment of Response to Treatment: WOMAC Physical Function Subscale and Subject Global Assessment of OA Condition
Subject Assessment | Day 14
  Subject Global Assessment of Response to Treatment: WOMAC Physical Function Subscale and Subject Global Assessment of OA Condition
Investigator Assessment | Day 3
  Investigator Global TCM Assessment of OA Condition: WOMAC Stiffness Subscale, Total WOMAC Index
Investigator Assessment | Day 7
  Investigator Global TCM Assessment of OA Condition: WOMAC Stiffness Subscale, Total WOMAC Index
Investigator Assessment | Day 14
  Investigator Global TCM Assessment of OA Condition: WOMAC Stiffness Subscale, Total WOMAC Index

CONTACTS AND LOCATIONS:
Overall Officials: Jackie (Yun) Mao, Study Director — Johnson & Johnson China
Locations (12):
- China (12):
  - Luoyang Orthopedic & Traumatologic Hospital of Henan Province, Luoyang, Hubei
  - Union Hospital affiliated to Tong Ji Medical College, Wuhan, Hubei
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - Jiang Su Province Hospital of TCM Hospital, Nanjing, Jiangsu
  - Su Zhou Chinese Medicine Hospital, Suzhou, Jiangsu
  - Wu Xi Chinese Medical Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Shan Xi TCM College, Xianyang, Shaanxi
  - Shanghai Chinese Medical Hospital, Shanghai, Shanghai Municipality
  - Shanghai Rui Jin Hospital, Shanghai, Shanghai Municipality
  - Shan Xi Provincial People's Hospital, Xi’an, Shanxi
  - Affiliated Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - 1st Affiliated Hospital of Tian Jin TCM College, Tianjin, Tianjin Municipality